CLINICAL TRIAL: NCT04260893
Title: A Prospective Study Assessing The Impact Of Tixel Treatment On Dry Eye Symptoms And Signs In Asian Patients With Dry Eye
Brief Title: Prospective Study To Assess The Safety And Effectiveness Of Tixel Treatment On Dry Eye Symptoms In Asian Patients
Acronym: DED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID19 adequate study monitoring wasn't possible by the Sponsor
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0734
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye Syndromes; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: All participants will undergo three sessions of treatments with the Investigation devise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tixel Treatment (Experimental): 3 Tixel treatment sessions, 2 weeks apart follow by 3 Follow up sessions
  Interventions: Device: Tixel

INTERVENTIONS:
Device: Tixel — Peri-Orbital fractional treatment on the Eye-Lid to assess the effect on Dry Eye symptoms
  Other Names: Fractional

SUMMARY:
Pilot study where effect of standard Tixel treatment as used for periorbital wrinkles would be assessed on Dry Eye Disease symptoms and signs in Asian Patients.

DETAILED DESCRIPTION:
Safety Assessment will be asses via AE/SAE reporting and Impact Assessment of the effect of the treatment on dry eye symptoms and signs through multiple

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years.
2. OSDI score of at least 23.
3. Noninvasive Tear film break up time (NIKBUT) ≤ 10 seconds.
4. No other eye or skin or immune problems.
5. Willing and able to provide written informed consent.
6. Willing to participate in all study activities and follow study instructions.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding.
2. Lesions in the periorbital area.
3. Acute severe blepharitis.
4. Acute conjunctivitis.
5. Concomitant anterior eye disease.
6. Has undergone outdoor/sunbed tanning during the last 4 weeks.
7. Is unwilling to follow the Tixel aftercare instructions after each of the three Tixel treatments.
8. Active Herpes Simplex or tendency for Herpes Simplex in the periorbital area (meaning the subject has had the condition previously).
9. Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
10. An impaired immune system condition or use of immunosuppressive medication.
11. Collagen disorders, keloid formation and/or abnormal wound healing.
12. Previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans for such treatment during the course of the Tixel treatments, or before complete healing of the treatments has occurred.
13. Has taken any medications (including via topical application), herbal treatment (oral or topic), food supplements or vitamins, which may cause fragile skin or impaired skin healing during the last 3 months.
14. Has used oral Isotretinoin (Accutane® or Roaccutan®) within 3 months prior to treatment.
15. History of bleeding coagulopathies or use of anticoagulants.
16. Tattoos or permanent makeup in the areas to be treated.
17. Burned skin, blistered skin, irritated skin, or sensitive skin in any of the areas to be treated.
18. Thread lifting of the area to be treated in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
SAFETY, number of AEs | 8 months
  Any safety related event during the study will be recorded and analysed
NIBUT in Seconds | 8 months
  Non-Invasive Break Up Time
Ocular Surface Disease Index Questionnaire | 8 months
  OSDI Score; 12 Questions; answers between 0-4; Total calculated. Higher score means worst Dry Eye Symptomes

SECONDARY OUTCOMES:
Topography mm D | 8 months
  Topography with K readings
Staining; Total Ocular Staining Score | 8 months
  Corneal staining fluorescein and conjunctival/lid margin staining lissamine green
Osmolarity mOsml/L | 8 months
  Osmolarity test with TearLab
Slit Lamp Exam; Normal, Abnormal | 8 months
  Multiple Slit Lamp tests
Meibography % | 8 months
  Calculate Meibography using IDRA device
Tear Meniscus Height mm | 8 months
  Tear Meniscus Height using IDRA device
Lid Wiper Epitheliopathy | 8 months
  Lid Wiper Epitheliopathy

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Shah, MD, Study Chair — University of Puthasastra; Mukesh Taneja, MD, Principal Investigator — University of Puthasastra
Locations (1):
- Khmer Sight Foundation Hospital, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No